CLINICAL TRIAL: NCT01743053
Title: A Pilot Trial of the Use of ReCell® Autologous Cell Harvesting Device for Venous Leg Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Avita Medical (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP003
Record Dates: First submitted 2012-11-29; First posted 2012-12-06 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Venous Leg Ulcers
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control: Standard Care (Other): The control group will receive standard care (debridement, cleansing) and Profore® multi-layer compression therapy (replacing the wound contact layer with Telfa™ Clear).
  Interventions: Other: Standard Care
- ReCell (Experimental): The ReCell group will receive ReCell in addition to standard care (debridement, cleansing) and Profore® multi-layer compression therapy (replacing the wound contact layer with Telfa Clear).
  Interventions: Device: Standard Care plus ReCell

INTERVENTIONS:
Device: Standard Care plus ReCell
  Arms: ReCell
Other: Standard Care
  Arms: Control: Standard Care

SUMMARY:
This is a prospective, randomised, open label, controlled pilot study to evaluate the safety and preliminary effectiveness of the ReCell Autologous Cell Harvesting Device (ReCell) for the management of chronic leg ulcers associated with venous insufficiency. Outcome will be compared between study participants receiving standard care (debridement, compression therapy) and participants receiving ReCell in addition to standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic venous leg ulcer (CEAP Clinical classification of 6)

   1. Confirmed, actively managed venous reflux
   2. No exposed tendon or bone
   3. Ulcer is >4 weeks in duration
   4. Ulcer surface area between 2cm2 and 80cm2
2. ABI ≥ 0.8
3. The patient is 18 years of age or older
4. The patient is willing to complete all follow-up evaluations required by the study protocol
5. The patient is able to abstain from any other treatment of the ulcer for the duration of the study, unless medically necessary
6. The patient agrees to abstain from enrolment in any other clinical trial for the duration of the study
7. The patient is able to read and understand instructions and give voluntary written informed consent
8. The patient is able and willing to follow the protocol requirements (including compression therapy)
9. Patients enrolling at any site in France must have an affiliation to a social security scheme

Exclusion Criteria:

1. Study treatment area has exposed bone or tendon
2. Poorly controlled diabetes
3. Arterial insufficiency (ABI < 0.8)
4. Pregnant/lactating females (self-reported or tested, per institutional requirements)
5. The patient has an active wound infection requiring antibiotic therapy
6. The patient has had a prior surgical treatment of the ulcer within the past 60 days
7. The patient has a life expectancy of 1-year or less
8. The patient has a severe dermatological disorder (e.g. severe psoriasis, epidermolysis bullosa, pyoderma gangrenosum).
9. The patient is unable to follow the protocol
10. The patient is taking, or has taken in the past 60 days, mycophenolate mofetil or >10mg of corticosteroids per day.
11. The patient has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives
12. The patient has a known hypersensitivity to trypsin or Compound Sodium Lactate for Irrigation (Hartmann's) solution.
13. The patient is a vulnerable or protected adult.
14. The patient is unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Wound healing | 12 weeks
  The primary objective of the study is to assess the difference in incidence of ulcer closure (investigator assessed as complete epithelialisation without drainage) between the ReCell group and the control group.

SECONDARY OUTCOMES:
Wounds characterization/Quality of Life | At each follow-up visit (1, 2, 4, 6, 8, 12, 24, 52 weeks)
  * Wound area
  * Wound volume
  * Pain
  * Recurrence
  * Health-related Quality of Life
Dressing Change | At each follow-up visit (1, 2, 4, 6, 8, 12, 24, 52 weeks) until healed
  - Dressing change

CONTACTS AND LOCATIONS:
Locations (7):
- Hôpital Lapeyronie, Montpellier, France
- United Kingdom (6):
  - Bradford Teaching Hospitals, Bradford
  - Cambridge University Hospitals - Addenbrooke's Hospital, Cambridge
  - Cardiff University, Cardiff
  - Doncaster and Bassetlaw Hospitals, Doncaster
  - The Leeds Teaching Hospitals - James's University Hospital, Leeds
  - University Hospital of South Manchester - Wythenshawe Hospital, Manchester